CLINICAL TRIAL: NCT04364984
Title: Effects of RAS Inhibitors (ARB, ACEi, DRI) in People With Hypertension 1-2 Stages on the Course of COVID-19 (BIRCOV Trial: ARB, ACEI, DRi Effects on COVID-19)
Brief Title: ARB, ACEi, DRi Effects on COVID-19 Course Disease
Acronym: BIRCOV
Status: Completed | Type: Observational
Sponsor: Medical Practice Prof D. Ivanov (Other)
Responsible Party: Sponsor
Other Study IDs: COVID20
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2021-08

CONDITIONS: Hypertension; COVID-19
Keywords: ACEi, ARB, DRI; Clinical features; CKD
MeSH Terms: conditions — Hypertension; COVID-19 | interventions — Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists; Renin Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ARB group: Hypertensive patients with COVID-19 who received ARBs
  Interventions: Drug: Angiotensin Receptor Blockers
- ACEi group: Hypertensive patients with COVID-19 who received ACEis
  Interventions: Drug: Angiotensin converting enzyme inhibitor
- DRi group: Hypertensive patients with COVID-19 who received direct renin inhibitor (DRis)
  Interventions: Drug: Direct renin inhibitor

INTERVENTIONS:
Drug: Angiotensin converting enzyme inhibitor — routine drug intake
  Other Names: no other drug as RAS inhibitor
  Groups: ACEi group
Drug: Angiotensin Receptor Blockers — routine drug intake
  Other Names: no other drug as RAS inhibitor
  Groups: ARB group
Drug: Direct renin inhibitor — routine drug intake
  Other Names: no other drug as RAS inhibitor
  Groups: DRi group

SUMMARY:
It is supposed to monitor hypertensive patients who are infected or have clinical manifestations of COVID-19 for 1 month after the onset of the disease. Three groups will be considered: 1. receiving ACE inhibitors 2. receiving ARBs 3. receiving DIR.

DETAILED DESCRIPTION:
POEM (Patient-Oriented Evidence that Matters) intervention is performed as an open prospective randomized two medical centres trial in subjects suffering from COVID-19 who have been receiving iRAS, either ACEi, ARB or DRi as basic antihypertensive therapy.

COVID-19 is confirmed by a PCR test, the disease follow-up is divided into 2 periods: up to 12 weeks and up to 24 weeks.

Primary Outcome Measure: BP was known one week before COVID-19 and is tested during the disease onset on weeks 2, 4, 12, 24. Secondary Outcome Measures are clinical features. Subanalysis in patients with CKD is additionally performed for those who have CKD.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive person, stage 1-2

Exclusion Criteria:

* Hypertensive subjects, stage 3, HF (NYHA) 3-4

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with proved COVID-19 and preliminary documented hypertension 1-2 stage on RASi at the onset and COVID-19 course during 3 weeks
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iryna Zavalna, MD, Study Chair — Nephrology clinic
Locations (1):
- Medical Practice Prof D.Ivanov, Kiev, Please Select, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 120 people with stage 1-2 hypertension have been screened. Study Population: patients with proved COVID-19 and preliminary stage 1-2 hypertension receiving iRAS at the onset of COVID-19.
  Minimum Age:18 Years, Maximum Age: 90 Years, Sex: All Inclusion Criteria: Hypertension, stage 1-2 with COVID-19. Exclusion Criteria: Hypertension, stage 3, HF (NYHA) 3-4
Groups:
- Group 1: ARB Group: 44 patients with COVID-19, hypertension 1-2 stages, who received ARB as main therapy for hypertension
- Group 2: iACE Group: 44 patients with COVID-19 and hypertension 1-2 stages, who received iACE as the main treatment for hypertensions
- Group 3: DRI Group: 31 patients with COVID-19, hypertension 1-2 stages, who received ARB as main therapy for hypertension
Period: Overall Study
Arm/Group | Group 1: ARB Group | Group 2: iACE Group | Group 3: DRI Group
Started | 37 | 44 | 31
Completed | 35 | 42 | 31
Not Completed | 2 | 2 | 0
Not completed — Death | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- ARB Group: Hypertensive patients with COVID-19 who received ARBs (valsartan 160-320 mg q.d. or olmesartan 20-40 mg q.d. or irbesartan 150-300 mg q.d. or candesartan 4-16 mg q.d.or losartan 50-100 mg q.d. in individual dosage) before and during COVID-19 for treatment of hypertension
- ACEi Group: Hypertensive patients with COVID-19 who received ACEis (enalapril 10-20 mg q.d. or ramipril 5-10 mg q.d. or lisinopril 10-20 mg q.d. or perindopril 5-10 mg q.d. in individual regime) before and during COVID-19 for treatment of hypertension
- DRi Group: Hypertensive patients with COVID-19 who received DRis (direct renin inhibitor rasilez in dosage 150-300 mg per day) before and during COVID-19 for treatment of hypertension
- Total: Total of all reporting groups
Arm/Group | ARB Group | ACEi Group | DRi Group | Total
Number analyzed (Participants) | 35 | 42 | 31 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 36 | 30 | 97
  >=65 years | 4 | 6 | 1 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] — documents and records
  years | 59 (1.8) | 55 (1.7) | 49 (1.4) | 55 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 9 | 48
  Male | 18 | 20 | 22 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Ukraine | 35 | 42 | 31 | 108

OUTCOME MEASURES:

1. Primary Outcome: Level of BP in mm Hg
Description: BP in patients one week before COVID-19 infection and 2, 4, 12, 24 weeks follow-up after COVID-19 onset
Time Frame: estimated at 2, 4, 12, 24 weeks after the start of COVID-19; data for 24 weeks are reported
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- DRi Group: Hypertensive patients with COVID-19 who received DRis
Arm/Group | ARB Group | ACEi Group | DRi Group
Number analyzed (Participants) | 35 | 42 | 31
mm Hg
  Systolic BP | 136 (1.1) | 138 (1.1) | 34 (1.4)
  Diastolic BP | 82 (1.2) | 83 (1.2) | 82 (1.2)

2. Secondary Outcome: Number of Patients With Fever Above 37.2 on COVID-19 Course
Description: the number of patients with hypertension who received RASi and has a fever (above 37.2C) separately on 2, 4 and 12 weeks follow-up
Time Frame: estimated at 2, 4, 12 weeks after the COVID-19 onset
Population: in the report, we document how many patients have a temperature above 37.2 on control data: 2, 4 and 12 weeks from COVID-19 onset
Measure: Count of Participants; unit: Participants
Arm/Group | ARB Group | ACEi Group | DRi Group
Number analyzed (Participants) | 35 | 42 | 31
Participants | 32 | 39 | 30

3. Secondary Outcome: Number of Patients With Cough in COVID-19 Course
Description: the absolute number of patients with hypertension on RASi who have had a cough at 2, 4 and 12 weeks from COVID-19 onset
Time Frame: on 2,4 and 12 week from COVID-19 onset
Measure: Count of Participants; unit: Participants
Arm/Group | ARB Group | ACEi Group | DRi Group
Number analyzed (Participants) | 35 | 42 | 31
Participants | 29 | 30 | 28

4. Secondary Outcome: Number of Patients With Throat Pain in COVID-19 Course
Description: the number of patients with hypertension on RASi with throat pain at 2, 4 and 12 weeks follow-up
Time Frame: estimated at 2, 4, 12 weeks after the COVID-19 onset
Measure: Count of Participants; unit: Participants
Arm/Group | ARB Group | ACEi Group | DRi Group
Number analyzed (Participants) | 35 | 42 | 31
Participants | 19 | 21 | 16

5. Secondary Outcome: Number of Patients With Diarrhea Inf COVID-19 Course
Description: the number of patients with hypertension on RASi with diarrhoea at 2, 4 and 12 weeks of follow-up
Time Frame: estimated at 2, 4, 12 weeks after the COVID-19 onset
Measure: Count of Participants; unit: Participants
Arm/Group | ARB Group | ACEi Group | DRi Group
Number analyzed (Participants) | 35 | 42 | 31
Participants | 3 | 4 | 1

6. Secondary Outcome: Number of Patients Who Need to Apply to Hospital in COVID-19 Course
Description: the number of patients with hypertension on RASi who need hospital and intensive care unit at 2, 4 and 12 weeks of follow-up
Time Frame: estimated at 2, 4, 12 weeks after the COVID-19 onset
Measure: Count of Participants; unit: Participants
Arm/Group | ARB Group | ACEi Group | DRi Group
Number analyzed (Participants) | 35 | 42 | 31
Participants | 2 | 2 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | ARB Group | ACEi Group | DRi Group
All-Cause Mortality (participants affected / at risk) | 2/35 | 2/42 | 0/31
Serious Adverse Events (participants affected / at risk) | 2/35 | 16/42 | 7/31
Other Adverse Events (participants affected / at risk) | 0/35 | 0/42 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARB Group (N=35) | ACEi Group (N=42) | DRi Group (N=31)
hypotension (Vascular disorders) | 2 (35) | 16 (42) | 7 (31) — hypotension as less than 110 mm Hg

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT04364984/Prot_SAP_000.pdf